CLINICAL TRIAL: NCT00371085
Title: Congestive Heart Failure Outreach Program (The COPE Study)
Brief Title: Congestive Heart Failure Outreach Program
Acronym: COPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Ross T. Tsuyuki, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EPICORE 2006-003
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Heart Failure
Keywords: heart failure; quality improvement; patient education; health care economics
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Video-based patient education on heart failure self care
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — Video-based educational program for heart failure focus on daily weights, medication taking, and salt restriction

SUMMARY:
Heart failure is a very common condition and is one of the main reasons people are admitted to hospital. There are many things people with heart failure can do to manage their condition at home. Unfortunately many people do not have enough information to do this and need to come back to the hospital because their heart failure got worse. This study will look at different ways to help people learn more about heart failure and how to manage their condition at home.

DETAILED DESCRIPTION:
Background:

Given the clinical and economic importance of heart failure (HF) widely applicable strategies to improve patient outcomes are needed. In Canada,1.4 million hospital days were associated with HF in the fiscal year 2000 and almost one-third of these were readmissions . The majority of acute precipitants of HF relate to poor self-care including excessive sodium and fluid intake, and nonadherence to medications. Data derived from the PaKSAC survey confirm that patients with HF have very poor knowledge of their condition and self-care recommendations.

Disease Management Programs for HF have been shown to improve clinical outcomes by providing intensive education and medical management. Due to the resource intensity of such programs, however, only a limited proportion of the population at risk is served. Clearly more practical educational interventions are needed.

Hypothesis:

An intervention consisting of a video-based educational program for patients with HF, focusing on 3 key steps (salt restriction, daily weights and medication adherence) will improve knowledge of self-care activities, and clinical and economic outcomes at 6 months of follow-up.

Design:

A multicentre randomized control trial comparing a simple, practical educational program for patients with heart failure to usual care. All patients will be assessed using the validated PaKSAC survey (Patient Knowledge of Self-Care Activities in Congestive Heart Failure) at baseline and at 6 months. Those randomized to the intervention will view a 22 minute educational video developed by our group that focuses on 3 key steps to self management. A booklet and series of 3 newsletters will also be provided to the intervention group. The primary outcome is the improvement in clinical outcomes at the end of the 6 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* patient in hospital or emergency room with symptomatic CHF confirmed by a physician.
* patient seen in an outpatient clinic with symptomatic CHF confirmed by a physician, AND hospitalized within the previous 6 months for heart failure.
* age greater than 18 years.

Exclusion Criteria:

* asymptomatic CHF
* life expectancy < 6 months
* receiving chronic hemodialysis or peritoneal dialysis
* unable to communicate (non-English speaking, intubated, etc)
* demented or a mental illness which precludes participation
* receives professional assistance for self-care activities including meals or medications (e.g. nursing home)
* previously enrolled in this study
* participation in another heart failure study, or
* declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2004-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Differences in clinical outcomes, as measured by cardiovascular hospitalizations and emergency room presentations, between video-based education and usual care groups. | 6 months

SECONDARY OUTCOMES:
Differences in all-cause hospitalizations between groups | 6 months
Differences in CHF-related hospitalizations between groups | 6 months
Differences in total number of in-hospital days between groups | 6 months
Change in CHF knowledge levels from the initial in-hospital patient contact to the end of the 6 month follow-up between the two groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, Pharm D, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital & others in Canada (contact PI), Edmonton, Alberta, Canada